CLINICAL TRIAL: NCT05821959
Title: A Trial of AAVAnc80-hOTOF Gene Therapy in Individuals With Sensorineural Hearing Loss Due to Otoferlin Gene Mutations
Brief Title: Gene Therapy Trial for Otoferlin Gene-mediated Hearing Loss
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akouos, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK-OTOF-101
Record Dates: First submitted 2023-02-08; First posted 2023-04-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: Otoferlin; Auditory neuropathy (AN); Deafness, autosomal recessive 9 (DFNB9); Hearing loss; Hearing loss, bilateral; Hearing loss, sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural; Deafness, Autosomal Recessive 9; Auditory neuropathy; Deafness; Hearing Loss; Hearing Loss, Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Cohort 1a and Cohort 1b (Experimental): Cohort 1a: Two participants aged 7 to 17 years old (inclusive) to receive intracochlear administration of AAVAnc80-hOTOF (dose level 1) in the study ear using a sterile, one-time use investigational medical device
  Cohort 1b: Up to six eligible participants will be enrolled to receive intracochlear administration of AAVAnc80-hOTOF (dose level 1) in the study ear using a sterile, one-time use investigational medical device; the first three participants will be at least two years of age at the time of AAVAnc80-hOTOF administration and the next three participants may be of any age
  Interventions: Combination Product: AAVAnc80-hOTOF via Akouos Delivery Device
- Cohort 2 (Experimental): Cohort 2: Up to six eligible participants will be enrolled to receive intracochlear administration of AAVAnc80-hOTOF (dose level 2) in the study ear using a sterile, one-time use investigational medical device; the first three participants will be at least two years of age at the time of AAVAnc80-hOTOF administration and the next three participants may be of any age
  Interventions: Combination Product: AAVAnc80-hOTOF via Akouos Delivery Device
- Bilateral Expansion (Experimental): Bilateral Expansion: up to eight eligible participants of any age, and no cochlear implants, may be eligible for enrollment into the Bilateral Expansion Cohort (simultaneous bilateral administration of AAVAnc80-hOTOF).
  Interventions: Combination Product: AAVAnc80-hOTOF via Akouos Delivery Device and Precision Delivery Mechanism

INTERVENTIONS:
Combination Product: AAVAnc80-hOTOF via Akouos Delivery Device — AAVAnc80-hOTOF is a sterile suspension intended to be administered via a one-time unilateral intracochlear administration using the Akouos Delivery Device.
  Arms: Cohort 1a and Cohort 1b; Cohort 2
Combination Product: AAVAnc80-hOTOF via Akouos Delivery Device and Precision Delivery Mechanism — AAVAnc80-hOTOF is a sterile suspension intended to be administered via a one-time bilateral intracochlear administration using the Akouos Delivery Device together with the Precision Delivery Mechanism.
  Arms: Bilateral Expansion

SUMMARY:
Part A of this trial will evaluate the safety and tolerability of a single surgical administration procedure in one or both ear(s) with one of two dose levels of AAVAnc80-hOTOF and will evaluate the Akouos Delivery Device, together with the Precision Delivery Mechanism, to safely achieve the intended product performance.

DETAILED DESCRIPTION:
The following two dose levels will be tested:

* Up to 4.1E11 total vg/cochlea
* Up to 8.1E11 total vg/cochlea

ELIGIBILITY:
Criteria for Inclusion:

1. Participants may be of any age, based on Cohort Criteria
2. At least two mutations in the otoferlin gene
3. Clinical presentation of Profound bilateral sensorineural hearing loss as assessed by ABR
4. Preserved distortion product otoacoustic emissions (DPOAEs)
5. Able and willing to comply with all study requirements, including willingness to participate in a separate long term follow-up study after completion of this trial

Criteria for Exclusion:

1. Persistent ear infections, anatomic or other abnormalities of the ear, and/or medical conditions that would contraindicate undergoing surgery, anesthesia, and/or administration of investigational gene therapy
2. Cochlear Implant(s) in the ear(s) to receive AAVAnc80-hOTOF
3. Prior participation in a clinical trial with an investigational drug, within six months prior to administration, or any prior participation in a gene therapy clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | through trial completion, approximately 1 year
  AEs with relationship to the investigational medicinal product and/or to the administration procedure (including the delivery system)

SECONDARY OUTCOMES:
Auditory Brainstem Response (ABR) Threshold | through trial completion, approximately 1 year
  Changes from baseline in ABR intensity threshold (decibels normal hearing level [dB nHL])
Performance of the Akouos Delivery Device and Precision Delivery Mechanism | through trial completion, approximately 1 year
  Performance based on the frequency of device deficiencies observed during delivery of AAVAnc80-hOTOF to the intracochlear space

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Reape, MD, Study Director — Akouos, Inc.
Locations (9):
- United States (6):
  - University of California, San Francisco Benioff Children's Hospital, San Francisco, California
  - University of Iowa, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt Bill Wilkerson Center, Nashville, Tennessee
- The Hospital for Sick Children Jaina.negandhi@sickkids.ca +1 (416) 813 6683, Toronto, Ontario, Canada
- National Taiwan University Hospital, Taipei, Taiwan
- University College London, London, United Kingdom, United Kingdom